CLINICAL TRIAL: NCT02724202
Title: A Pilot, Feasibility Study of Curcumin in Combination With 5FU for Patients With 5FU-Resistant Metastatic Colon Cancer
Brief Title: Curcumin in Combination With 5FU for Colon Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI-Initiated study; PI requested closure
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 014-143
Record Dates: First submitted 2016-03-16; First posted 2016-03-31 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colon Cancer
Keywords: Curcumin; 5FU; 5-fluorouracil; Adracil; 5FU Resistant; Metastatic Colon Cancer; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Curcumin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): All subjects will receive induction oral curcumin 500 mg twice per day for 2 weeks. Patients will continue on curcumin at same dose for an additional 6 weeks while being treated with 3 cycles of 5FU.
  Interventions: Drug: Curcumin; Drug: 5-flurorouracil

INTERVENTIONS:
Drug: Curcumin — Curcumin is supplied as soft-gel capsule. It is a micronized rhizome extract containing phospholipids and 500mg of pure curcuminoids (95% curcumin, 5% desmethoxycurcumin) suspended in turmeric essential oil.
  Other Names: BCM-95
Drug: 5-flurorouracil — Fluorouracil is an anti-cancer (antineoplastic or cytotoxic) chemotherapy drug. Fluorouracil is classified as an antimetabolite.
  Other Names: 5FU; Adracil

SUMMARY:
The purpose of this study is to test the safety and find the response rate of combining the dietary supplement, curcumin, with the standard of care, FDA-approved chemotherapy drug 5-fluorouracil (5FU, Adracil) and see what effects (good and bad) that the combined treatments have on colon cancer.

DETAILED DESCRIPTION:
Confirm clinical safety and identify clinical response rate of combination treatment with curcumin and 5FU in chemorefractory CRC patients. To determine whether curcumin administration induces systemic alterations in inflammatory and epigenetic biomarkers in patients with chemoresistant metastatic colorectal cancer (CRC). To correlate altered biomarker findings with clinical response according to RECIST V1.1 and survival criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older, at the time of signing the informed consent.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Histologically or cytologically confirmed diagnosis of metastatic colorectal cancer that is not response to standard 5FU based therapies.
* Performance Status (PS) score of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain oral medication.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 mili-internation unit (MIU)/ml and estradiol <40 pg/ml (140pmol/L) is confirmatory
* Child-bearing potential and agrees to use a contraception method of abstinence, intrauterine device (IUD), barrier methods or birth control pills prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point and until three months after the last dose of the study medication.
* Male subjects must agree to use a method of contraception. This criterion must be followed from the time of the first dose of study medication until three months after the last dose of study medication.
* Adequate organ system function defined as follows:

System Laboratory Values Hematologic Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L Hemoglobin ≥ 9.5 g/dL Platelets ≥ 75 x 10^9/L For subjects not on warfarin-based anticoagulants: Prothrombin time/International normalized ratio (PT/INR) and partial thromboplastin time (PTT) ≤ 1.1x upper limit of normal (ULN) INR (subjects on warfarin-based anticoagulant): 2-3 x ULN Hepatic Total bilirubin ≤ 1.5x ULN (isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) Aspartate aminotransferase (AST) and alanine transaminase (ALT) 1 ≤ 1.5x ULN Albumin ≥ 2.5 g/dL Renal Creatinine ≤ ULN; or Calculated creatinine clearance2 ≥ 50 mL/min; or Metabolic Fasting Serum Glucose < 250 mg/dL Cardiac Left Ventricular Ejection fraction (LVEF) ≥ lower limit of normal (LLN) by echocardiogram (ECHO) Blood pressure Systolic < 160 mm Hg and Diastolic < 100 mm Hg.

1. If liver metastases are present, AST and ALT ≤ 2.5x ULN is permitted
2. As calculated by Cockcroft-Gault formula.

Exclusion Criteria:

* Chemotherapy, radiotherapy, immunotherapy, or other anti-cancer therapy including investigational drugs within 28 days or 5 half-lives, whichever is shorter prior to the first dose of any one of the investigational drugs described in this study.
* Unresolved toxicity by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE V4) of > Grade 1 from previous anti-cancer therapy.
* Presence of active GI disease or other condition that could affect gastrointestinal absorption (malabsorption syndrome) or predispose a subject to GI ulceration.
* Evidence of mucosal or internal bleeding
* Any major surgery within the last four weeks
* Uncontrolled diabetes mellitus
* Any malignancy related to human immunodeficiency virus (HIV), known history of HIV, history of known Hepatitis B virus (HBV) surface antigen positivity (subjects with documented laboratory evidence of HBV clearance may be enrolled) or positive Hepatitis C virus (HCV) antibody.
* Known active infection requiring parenteral or oral anti-infective treatment.
* Subjects with brain metastases are excluded if their brain metastases are:
* Symptomatic
* Treated (surgery, radiation therapy) but not clinically and radiographically stable one month after therapy (as assessed by at least 2 distinct contrast enhanced MRI or CT scans over at least a one month period), or
* Asymptomatic and untreated but > 1 cm in the longest dimension
* History or evidence of current clinically significant uncontrolled arrhythmias.
* Subjects with controlled atrial fibrillation for >1 month prior to study Day 1 are eligible.
* History of acute coronary syndromes (including unstable angina), myocardial infarction, coronary angioplasty, or stenting or bypass grafting within six months of screening.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Any serious or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject's safety or providing informed consent.
* Known immediate or delayed hypersensitivity to any of the components of the study treatment(s).
* Evidence of severe or uncontrolled systemic diseases (unstable or uncompensated respiratory, hepatic, renal, or cardiac disease, including unstable hypertension).
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety using curcumin in patients with metastatic colon cancer; where toxicities will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. | 12 weeks
  Events will be recorded from the time of informed consent signature through the 30 days following the last study treatment.

SECONDARY OUTCOMES:
Overall Response | 12 months
  Recorded from the start of the treatment until disease progression/recurrence. The patient's best response assignment will depend on the finding of target and non-target disease and will also take into consideration the appearance of new lesions.
Evidence of altered biomarker status (circulating DNA methylation status, miRNA profile) at 8 weeks post-treatment according to RECIST version 1.1 and survival criteria. | Baseline, Week 2, Week 8
  Blood will be collected at baseline, after completing one cycle of curcumin treatment (2 weeks), and after completing three 2 week-cycles of 5FU (6 weeks) for inflammatory and epigenetic chemoresponsive biomarker profiling.
Duration of response | 12 months
Duration of progression free survival | 12 months
Duration of overall survival | 12 months
Duration of Quality of Life | Baseline, 12 months
  All subjects will complete the quality of life survey at Baseline, 5FU treatment visits and follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: John Preskitt, MD, Principal Investigator — Baylor University Medical Center/Texas Oncology, PA
Locations (1):
- Baylor Charles A. Sammons Cancer Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes